CLINICAL TRIAL: NCT03543163
Title: The Evaluation of Recession Depth After Treating Miller Class I and II Gingival Recession Using Non- Pedicled Buccal Fat Pad Graft as Compared to Subepithelial Connective Tissue Graft. A Randomized Controlled Clinical Trial
Brief Title: Treatment of Miller Class I and II Gingival Recession Using Non- Pedicled Buccal Fat Pad Graft as Compared to Subepithelial Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alia Emad Mohammed, associate lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-05-15
Record Dates: First submitted 2018-05-19; First posted 2018-06-01 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Gingival Recession
Keywords: buccal fat pad graft; sub-epithelial connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: * Blinding of the participants is not applicable.
  * Blinding of the operator is not applicable.
  * Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subepithelial connective tissue graft (Active Comparator): Subepithelial Connective Tissue graft from the hard palate with Coronally Advanced flap at the site of gingival recession.
  Interventions: Procedure: sub-epithelial connective tissue graft
- non pedicled buccal fat pad graft (Experimental): Non- Pedicled Buccal Fat Pad with Coronally Advanced flap at the site of gingival recession
  Interventions: Procedure: Non- Pedicled Buccal Fat Pad with Coronally Advanced flap

INTERVENTIONS:
Procedure: Non- Pedicled Buccal Fat Pad with Coronally Advanced flap — A horizontal incision of 1.5cm in long will be made at the bottom of the vestibule with the #15 blade in the region of maxillary first and second molars, depending on side of the recipient site. A curved hemostat will be used in the blunt dissection through the buccinators muscle to temporarily reposition and loose the surrounding fascia which will allow the buccal fat pad to be exposed in the oral cavity. A portion of adipose tissue equals to the required graft size will be excised with the microsurgical scissors. The grafting material will be placed on a saline-soaked gauze until its transfer to the recipient site. Finally, the patient's check will be compressed, in order to promote the closure of the wound edges then immediately close the donor site with simple 5.0 silk thread interrupted sutures
  Arms: non pedicled buccal fat pad graft
Procedure: sub-epithelial connective tissue graft — a sub- epithelial connective tissue graft is harvested from the hard palate is used to treat area with gingival recession
  Arms: subepithelial connective tissue graft

SUMMARY:
This randomized controlled single blinded parallel clinical trial is held to monitor if the use of the non pedicled buccal fat pad graft will result in post operative pain as a primary outcome compared to that occurs with the use of the sub epithelial connective tissue graft in treating Miller Class I and Class II gingival recession

ELIGIBILITY:
Inclusion Criteria:

1. Patients are systemically healthy based on questionnaire dental modification of Cornell index.
2. Patients are periodontally healthy with no contraindication for periodontal surgery.
3. All patients are not using any kind of medications that could interfere with the health of gingiva or periodontal tissues.
4. O'Leary index is less than 10% ( the surgical therapy is not initiated until the patient reaches the 10% level or less of plaque accumulation)
5. Buccal recession defects are classified as Miller Class I or II.
6. Presence of identifiable CEJ.
7. The papilla fill the interdental spaces as far as the contact area
8. Clinical indication and/or patient request for recession coverage.

Exclusion Criteria:

1. Miller Class III or IV recession defects
2. Pregnant female.
3. Smokers as smoking is contraindicated for any plastic periodontal surgery
4. Patients with special needs or with any mental problems.
5. Patients undergoing radiotherapy
6. Teeth with carious or non-carious lesion or cervical restorations
7. Rotated teeth and tooth extrusion with or without occlusal abrasion
8. Patient undergone any prior periodontal surgery in the relevant region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recession Depth | 6 months
  Measured from the CEJ to the most apical extension of the gingival margin using the UNC-15 periodontal probe and measured in mm unit

SECONDARY OUTCOMES:
Thickness of keratinized tissue | 6 months
  Evaluation of the gingival thickness by trans-gingival piercing using an anesthetic needle with a silicon stopper inserted perpendicular to the mucosal surface with light pressure until touching a hard surface and the silicon disk in a tight contact with soft tissue surface. This measurement should be taken 1.5 mm apical from the gingival margin. Then the correct position of the disk is fixed with a drop of cyanoacrylic adhesive after careful removal of the needle. The penetration depth is measured by an accurate caliper
Post-operative pain | 2 weeks
  Visual Analogue Scale (VAS) with numbers from 0 to 100 ('no pain' to 'worst pain